CLINICAL TRIAL: NCT00066001
Title: The Effect of Systemically Administered Metronidazole Alone and in Combination With Professional Supragingival Plaque Removal on Plaque Composition
Brief Title: Microbial Associations in Periodontal Health and Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Forsyth Institute (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Ann D. Haffajee/PI/Chair Department of Periodontology/Senior Member of the Staff, The Forsyth Instititute
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDCR-12108; R01DE012108 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Periodontitis; Periodontal Diseases
MeSH Terms: conditions — Periodontitis; Periodontal Diseases | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1, 2, 3, 4 (Placebo Comparator): The 4 arms of the study are based on the treatment groups: 1. scaling and root planing alone (SRP); 2. SRP plus repeated professional supragingival plaque removal; 3. SRP + systemically administered metronidazole; 4. SRP + repeated professional supragingival plaque removal + systemically administered metronidazole.
  Interventions: Drug: metronidazole

INTERVENTIONS:
Drug: metronidazole — antibiotic that is particularly effective against Gram negative bacterial species

SUMMARY:
The purpose of this study is to determine the clinical and microbiological effects of systemically administered metronidazole alone or in combination with professional plaque removal on periodontally diseased patients.

DETAILED DESCRIPTION:
Major goals of periodontal research are to differentiate pathogenic from host compatible plaque microbiotas and to optimize treatments to convert the former to the latter. To this end, in the previous award period the composition of supra and subgingival plaques, the associations among species both within and between supra and subgingival plaques, and differences between plaques from healthy and diseased individuals were determined. One major finding was the frequent detection of anaerobic periodontal pathogens at low numbers in supragingival plaque of periodontally diseased and to a lesser extent healthy subjects. Weekly professional supragingival plaque removal for 3 months in 18 periodontitis subjects demonstrated astonishing reductions in the subgingival microbiota which were maintained for 9 months after cessation of the professional program. The composition of the microbiota at 12 months in these subjects was similar to that found in periodontal health. In another of our studies, systemically administered metronidazole produced similar effects. Thus, in SA1 a 2 year randomized clinical trial will be performed comparing the effects of 1) SRP alone or in combination with 2) weekly professional supragingival plaque removal, 3) systemically administered metronidazole or 4) a combination of the 2 on clinical parameters and supra and subgingival plaque composition. 200 periodontitis patients will receive SRP under local anaesthesia and will be randomly assigned to the 4 treatment groups. All subjects will be evaluated clinically and for supra and subgingival plaque composition at 2 weeks, 3, 6, 12, 18 and 24 months. Supra and subgingival plaque samples will be taken separately from the mesial aspect of each tooth and evaluated individually for their content of 40 bacterial species using checkerboard DNA-DNA hybridization providing over 3.6 million bacterial counts. The results will determine if the beneficial effect of the individual therapies persist beyond one year and whether combined treatment produces even greater benefit to the patient.

ELIGIBILITY:
Inclusion:

* > 35 years of age
* > 20 teeth
* > 5% sites (approx. 8 sites) with pocket depth > 4 mm and / or 5% sites with attachment level > 4 mm

Exclusion:

* > 50% of sites with pocket depth or attachment level > 4 mm
* Pregnancy or lactation
* Periodontal or antibiotic therapy in the previous 12 months
* Any systemic condition which might influence the course of periodontal disease or treatment (e.g. diabetes, AIDS)
* Any systemic condition which requires antibiotic coverage for routine periodontal procedures (e.g. heart conditions, joint replacements etc.)
* Any known allergy to metronidazole

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2002-12; Primary Completion 2007-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in mean attachment level | Baseline, 3, 6 12 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann Haffajee, Principal Investigator — Boston, MA
Locations (1):
- Department of Periodontology, The Forsyth Institute, Boston, Massachusetts, United States